CLINICAL TRIAL: NCT03187002
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Control During First Trimester Abortion: A Blinded Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Control During First Trimester Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-41589
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Abortion in First Trimester
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcutaneous electrical nerve stimulation (TENS) (Experimental): Transcutaneous electrical nerve stimulation (TENS)
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS); Other: SHAM: Moderate IV Sedation
- Moderate IV Sedation (Active Comparator): Fentanyl, versed
  Interventions: Drug: Moderate IV Sedation; Other: SHAM: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve-stimulation (TENS) is a nonpharmacologic means of pain control that delivers electrical currents through the skin. These pulses of electrical current reduce pain by peripheral and central mechanisms, TENS actives descending inhibitory systems in the central nervous system to reduce sensitivity to pain (hypoalgesia). Assessment of previous TENS research identifies intensity as a critical factor in efficacy-documenting high intensity as the best means of pain control, as the higher pulse allows for deeper tissue afferents to be activated. TENS has been researched in a number of settings as pain control, including cancer pain, lower back pain, labor, and a range of gynecologic procedures and disorders.
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Drug: Moderate IV Sedation — IV sedation with fentanyl and versed
  Arms: Moderate IV Sedation
Other: SHAM: Transcutaneous electrical nerve stimulation (TENS) — Sham Transcutaneous electrical nerve stimulation (TENS) to ensure blinding
  Arms: Moderate IV Sedation
Other: SHAM: Moderate IV Sedation — Sham IV to ensure blinding
  Arms: Transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
High-frequency, high-intensity transcutaneous electrical nerve-stimulation (TENS) is an inexpensive and non-invasive pain control approach. TENS, pulsating electrical currents that activate underlying nerves, does not have drug interactions or risk of overdose. Cochrane review of TENS for acute pain found inconclusive evidence. One previous abortion trial comparing TENS to IV sedation only looked at pain control in the recovery room. The investigators propose a randomized controlled trial comparing TENS to IV sedation (in conjunction with local anesthesia) among women presenting for first-trimester surgical abortion. Primary outcome will be perceived pain by Visual Analogue Scale (VAS) during aspiration.

ELIGIBILITY:
Inclusion criteria:

* Presenting for surgical abortion
* Gestational age <12 weeks
* < 18 years of age
* Agrees to be randomized

Exclusion criteria:

* Allergy to study medications (lidocaine, fentanyl, midazolam)
* > 18 years of age
* Fetal demise
* Pre-procedure use of misoprostol
* No means of transportation following procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, Principal Investigator — Stanford University
Locations (1):
- Planned Parenthood Mar Monte, San Jose, California, United States

REFERENCES:
- [Derived] Lerma K, Goldthwaite LM, Blumenthal PD, Shaw KA. Transcutaneous Electrical Nerve Stimulation for Pain Management of Aspiration Abortion up to 83 Days of Gestation: A Randomized Controlled Trial. Obstet Gynecol. 2021 Sep 1;138(3):417-425. doi: 10.1097/AOG.0000000000004502. PMID 34352845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment occurred at the Planned Parenthood site.
Period: Overall Study
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Started | 55 | 54
Completed | 55 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.5) | 28 (6) | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 47
  Not Hispanic or Latino | 32 | 25 | 57
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 4 | 4 | 8
  White | 21 | 17 | 38
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109
Gestational Age [Median (Full Range); unit: days] — Measured by ultrasound on day of enrollment and procedure
  days | 53 [36 to 82] | 58 [35 to 82] | 55 [35 to 82]

OUTCOME MEASURES:

1. Primary Outcome: Aspiration Pain
Description: Pain with aspiration, assessed by visual analogue scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure at the time of aspiration (up to 30 seconds)
Population: 9 participants required rescue medication (IV sedation with fentanyl and versed) during the procedure in the TENS group and were excluded from per-protocol analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 73 [13 to 97] | 66 [0 to 99]

2. Secondary Outcome: Speculum Placement Pain
Description: Pain with speculum placement, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure (up to 30 seconds)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 27 [0 to 97] | 17.5 [0 to 98]

3. Secondary Outcome: Tenaculum Placement Pain
Description: Pain at time of tenaculum placement, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure (up to 30 seconds)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 34.5 [0 to 82] | 23.5 [0 to 72]

4. Secondary Outcome: Paracervical Block Pain
Description: Pain with paracervical block, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure (up to 30 seconds)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 48.5 [0 to 87] | 34.5 [3 to 81]

5. Secondary Outcome: Manual Cervical Dilation Pain
Description: Pain with manual cervical dilation, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure (up to 30 seconds)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 67 [11 to 94] | 56 [0 to 99]

6. Secondary Outcome: Speculum Removal Pain
Description: Pain with speculum removal, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intraoperative, collected during procedure (up to 30 seconds)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
units on a scale | 38.5 [0 to 83] | 23 [0 to 94]

7. Secondary Outcome: Total Procedure Time
Description: Time from speculum placement to speculum removal, measured in minutes
Time Frame: Intraoperative, collected during procedure (up to 20 minutes)
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
Number analyzed (Participants) | 46 | 54
minutes | 7 [3.5 to 16.5] | 6.4 [3.3 to 16.4]

ADVERSE EVENTS:
Time Frame: Up to 4 hours
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Moderate IV Sedation
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03187002/Prot_SAP_000.pdf